CLINICAL TRIAL: NCT04661046
Title: Study on the Correlation Between Gene Mutation and TCM Syndrome Types in Metastatic Colorectal Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: SHSLCZDZK 03701
Record Dates: First submitted 2020-11-20; First posted 2020-12-09 (Actual); Last update posted 2020-12-09 (Actual); Status verified 2020-11

CONDITIONS: Gene Mutation-Related Cancer; Traditional Chinese Medicine
MeSH Terms: interventions — Medicine, Chinese Traditional

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TCM Syndrome Types (Experimental): Traditional Chinese Medicine
  Interventions: Drug: Traditional Chinese Medicine

INTERVENTIONS:
Drug: Traditional Chinese Medicine — Chinese medicine prescription
  Other Names: TCM

SUMMARY:
To explore the correlation between gene mutations of metastatic colorectal cancer and TCM syndrome types based on Second-generation sequencing technology.

ELIGIBILITY:
Inclusion Criteria:

1. A clear pathological diagnosis is a patient with colorectal cancer;
2. Have complete TNM staging information;
3. There is a clear diagnosis of the location and time of metastasis;
4. Age ≥18 years old, ≤80 years old, male or female;
5. There is a clear time for the first treatment with Chinese medicine;
6. Patients who can receive long-term follow-up. -

Exclusion Criteria:

1. Patients with colorectal cancer diagnosed pathologically as adenosquamous carcinoma, squamous cell carcinoma, carcinoid, small cell carcinoma, malignant lymphoma, etc.;
2. Patients with double cancer, multiple or metastatic colorectal cancer;
3. Combined with severe acute and chronic diseases that may affect treatment and prognosis, such as myocardial infarction, stroke, severe renal insufficiency and mental illness;-

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-11-30 (Estimated); Primary Completion 2022-08-31 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | 2 years
  OS
Progression Free Survival | 2 years
  PFS

IPD SHARING:
Plan to Share IPD: Undecided